CLINICAL TRIAL: NCT04840940
Title: Presepsin as an Early Biomarker for Ventilator-associated Pneumonia (VAP) Diagnosis in COVID-19 Patients: a Prospective Double Blind Observational Study
Brief Title: Presepsin Biomarker for Ventilator-associated Pneumonia Diagnosis in COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Pietro Caironi, Director, Department of Anesthesia and Critical Care, San Luigi Gonzaga Hospital
Other Study IDs: MACOSX
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Ventilator Associated Pneumonia; Covid19
Keywords: Presepsin; VAP; Mechanical ventilation; COVID-19; Ventilator associated pneumonia; Sars-Cov-2
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Presepsin serum level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is observational and double blind. It evaluates the validity of presepsin (a serum biomarker of bacterial infections) as early biomarker of Ventilator Associated Pneumonia. It will be measured at day 0 (ICU admission) and every 48 hours in every patient with Sars-Cov 2 interstitial pneumonia requiring invasive mechanical ventilation (see inclusion ad exclusion criteria) until Day 30, ICU discharge or ICU death. There will be no change in clinical practice and in pneumonia diagnosis. We will examine how the elevation of presepsin level could be an early marker of ventilator associated pneumonia or a marker of bacterial pneumonia at ICU admission, before the microbiological results or clinical diagnosis.

DETAILED DESCRIPTION:
This study will be a single center, double blind observational study.

Measurements of presepsin blood level will be performed in all patients with interstitial Sars-Cov-2 pneumonia admitted to ICU, at the time of the start of invasive mechanical ventilation and every 48 hours for the first 30 days of ICU stay. Surveillance respiratory samples (endotracheal aspiration) will be performed according to clinical practice (at ICU admission and every Mondays and Thursdays in all patients undergoing invasive mechanical ventilation).

In all patients admitted to ICU with invasive mechanically ventilation, a bronchoalveolar lavage with rapid microbiological method (film array for the research of the main respiratory pathogens) will be performed, according to common clinical practice.

VAP diagnosis will be made based upon the evidence of new lung infiltrates (chest radiography or chest computed tomography) in association with the presence of a pathogen isolated in the non-invasive respiratory sample with semi-quantitative method, according to IDSA and American Thoracic Society guidelines, as well as the presence of other sign of infection (fever, leukocytosis, worsening of oxygenation).

The attending physician in charge of the patient enrolled, clinically making the diagnosis of VAP will be blinded of presepsin levels. As a consequence, during the study period, no variation of the clinical practice applied will be performed, and no influence on the care provided to patients included will be determined by the measurement of plasma presepsin.

In the current study, we aim to answer to the following questions:

* Does a high level of plasma presepsin in patients with a Sars Cov 2 interstitial pneumonia at the time of ICU admission predict the presence of a bacterial respiratory co-infection?
* Do presepsin levels early predict the occurrence of VAP in patients with COVID-19 disease?
* Does such variation become evident at the time of VAC, therefore anticipating the diagnosis of IVAC? The latter issue might be particularly important in order to commence antibiotic therapy earlier than the diagnosis of IVAC.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with Sars Cov 2 interstitial pneumonia requiring invasive mechanical ventilation

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Chronic renal failure stage III or more
* End stage liver disease
* Patients already present in the ICU at the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring invasive mechanical ventilation for Sars-Cov 2 interstitial pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-12-21 (Estimated); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
To evaluate daily variations of presepsin levels as an early marker of VAP in COVID 19 patients | Time from ICU admission to day 30 or to ICU discharge or to ICU death
  Circulating presepsin levels every other day (from day 0 to day 30)

SECONDARY OUTCOMES:
To evaluate whether presepsin level can predict the presence of a bacterial respiratory co-infection at the time of ICU admission in patient with Sars-CoV-2 interstitial pneumonia | Time from ICU admission to day 2
  Circulating presepsin levels every other day (from day 0 to day 2)
To evaluate the role of circulating presepsin time course during the treatment of VAP as a clinical marker of the adequacy of the antibiotic therapy applied | Time from ICU admission to day 30 or to ICU discharge or to ICU death
  Circulating presepsin levels every other day (from day 0 to day 30)
To evaluate whether plasma levels of presepsin may distinguish the presence of VAP versus VAT (ventilator-associated tracheobronchitis). | Time from ICU admission to day 30 or to ICU discharge or to ICU death
  Circulating presepsin levels every other day (from day 0 to day 30)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Caironi, Principal Investigator — San Luigi Gonzaga Hospital; Guido Bussone, Principal Investigator — San Luigi Gonzaga Hospital
Locations (1):
- SCDU Anestesia e Rianimazione, AOU San Luigi Gonzaga, Orbassano, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Result] Melsen WG, Rovers MM, Groenwold RH, Bergmans DC, Camus C, Bauer TT, Hanisch EW, Klarin B, Koeman M, Krueger WA, Lacherade JC, Lorente L, Memish ZA, Morrow LE, Nardi G, van Nieuwenhoven CA, O'Keefe GE, Nakos G, Scannapieco FA, Seguin P, Staudinger T, Topeli A, Ferrer M, Bonten MJ. Attributable mortality of ventilator-associated pneumonia: a meta-analysis of individual patient data from randomised prevention studies. Lancet Infect Dis. 2013 Aug;13(8):665-71. doi: 10.1016/S1473-3099(13)70081-1. Epub 2013 Apr 25. PMID 23622939
- [Result] Magill SS, Klompas M, Balk R, Burns SM, Deutschman CS, Diekema D, Fridkin S, Greene L, Guh A, Gutterman D, Hammer B, Henderson D, Hess D, Hill NS, Horan T, Kollef M, Levy M, Septimus E, VanAntwerpen C, Wright D, Lipsett P. Developing a new, national approach to surveillance for ventilator-associated events*. Crit Care Med. 2013 Nov;41(11):2467-75. doi: 10.1097/CCM.0b013e3182a262db. PMID 24162674
- [Result] Erb CT, Patel B, Orr JE, Bice T, Richards JB, Metersky ML, Wilson KC, Thomson CC. Management of Adults with Hospital-acquired and Ventilator-associated Pneumonia. Ann Am Thorac Soc. 2016 Dec;13(12):2258-2260. doi: 10.1513/AnnalsATS.201608-641CME. No abstract available. PMID 27925784
- [Result] Berton DC, Kalil AC, Teixeira PJ. Quantitative versus qualitative cultures of respiratory secretions for clinical outcomes in patients with ventilator-associated pneumonia. Cochrane Database Syst Rev. 2012 Jan 18;1:CD006482. doi: 10.1002/14651858.CD006482.pub3. PMID 22258968
- [Result] Fagon JY. Biological markers and diagnosis of ventilator-associated pneumonia. Crit Care. 2011;15(2):130. doi: 10.1186/cc10050. Epub 2011 Mar 9. PMID 21418551
- [Result] Luyt CE, Combes A, Reynaud C, Hekimian G, Nieszkowska A, Tonnellier M, Aubry A, Trouillet JL, Bernard M, Chastre J. Usefulness of procalcitonin for the diagnosis of ventilator-associated pneumonia. Intensive Care Med. 2008 Aug;34(8):1434-40. doi: 10.1007/s00134-008-1112-x. Epub 2008 Apr 18. PMID 18421435
- [Result] Luyt CE, Guerin V, Combes A, Trouillet JL, Ayed SB, Bernard M, Gibert C, Chastre J. Procalcitonin kinetics as a prognostic marker of ventilator-associated pneumonia. Am J Respir Crit Care Med. 2005 Jan 1;171(1):48-53. doi: 10.1164/rccm.200406-746OC. Epub 2004 Sep 24. PMID 15447947
- [Result] COVID-ICU Group on behalf of the REVA Network and the COVID-ICU Investigators. Clinical characteristics and day-90 outcomes of 4244 critically ill adults with COVID-19: a prospective cohort study. Intensive Care Med. 2021 Jan;47(1):60-73. doi: 10.1007/s00134-020-06294-x. Epub 2020 Oct 29. PMID 33211135
- [Result] Mussap M, Noto A, Fravega M, Fanos V. Soluble CD14 subtype presepsin (sCD14-ST) and lipopolysaccharide binding protein (LBP) in neonatal sepsis: new clinical and analytical perspectives for two old biomarkers. J Matern Fetal Neonatal Med. 2011 Oct;24 Suppl 2:12-4. doi: 10.3109/14767058.2011.601923. PMID 21740312
- [Result] Okamura Y, Yokoi H. Development of a point-of-care assay system for measurement of presepsin (sCD14-ST). Clin Chim Acta. 2011 Nov 20;412(23-24):2157-61. doi: 10.1016/j.cca.2011.07.024. Epub 2011 Aug 3. PMID 21839732
- [Result] Wu CC, Lan HM, Han ST, Chaou CH, Yeh CF, Liu SH, Li CH, Blaney GN 3rd, Liu ZY, Chen KF. Comparison of diagnostic accuracy in sepsis between presepsin, procalcitonin, and C-reactive protein: a systematic review and meta-analysis. Ann Intensive Care. 2017 Sep 6;7(1):91. doi: 10.1186/s13613-017-0316-z. PMID 28875483
- [Result] Masson S, Caironi P, Fanizza C, Thomae R, Bernasconi R, Noto A, Oggioni R, Pasetti GS, Romero M, Tognoni G, Latini R, Gattinoni L. Circulating presepsin (soluble CD14 subtype) as a marker of host response in patients with severe sepsis or septic shock: data from the multicenter, randomized ALBIOS trial. Intensive Care Med. 2015 Jan;41(1):12-20. doi: 10.1007/s00134-014-3514-2. Epub 2014 Oct 16. PMID 25319385
- [Result] Masson S, Caironi P, Spanuth E, Thomae R, Panigada M, Sangiorgi G, Fumagalli R, Mauri T, Isgro S, Fanizza C, Romero M, Tognoni G, Latini R, Gattinoni L; ALBIOS Study Investigators. Presepsin (soluble CD14 subtype) and procalcitonin levels for mortality prediction in sepsis: data from the Albumin Italian Outcome Sepsis trial. Crit Care. 2014 Jan 7;18(1):R6. doi: 10.1186/cc13183. PMID 24393424
- [Result] Klouche K, Cristol JP, Devin J, Gilles V, Kuster N, Larcher R, Amigues L, Corne P, Jonquet O, Dupuy AM. Diagnostic and prognostic value of soluble CD14 subtype (Presepsin) for sepsis and community-acquired pneumonia in ICU patients. Ann Intensive Care. 2016 Dec;6(1):59. doi: 10.1186/s13613-016-0160-6. Epub 2016 Jul 7. PMID 27389015
- [Result] Zaninotto M, Mion MM, Cosma C, Rinaldi D, Plebani M. Presepsin in risk stratification of SARS-CoV-2 patients. Clin Chim Acta. 2020 Aug;507:161-163. doi: 10.1016/j.cca.2020.04.020. Epub 2020 Apr 22. PMID 32333860
- [Result] Fukada A, Kitagawa Y, Matsuoka M, Sakai J, Imai K, Tarumoto N, Orihara Y, Kawamura R, Takeuchi S, Maesaki S, Maeda T. Presepsin as a predictive biomarker of severity in COVID-19: A case series. J Med Virol. 2021 Jan;93(1):99-101. doi: 10.1002/jmv.26164. Epub 2020 Jun 24. No abstract available. PMID 32530491
- [Result] Schirinzi A, Cazzolla AP, Lovero R, Lo Muzio L, Testa NF, Ciavarella D, Palmieri G, Pozzessere P, Procacci V, Di Serio F, Santacroce L. New Insights in Laboratory Testing for COVID-19 Patients: Looking for the Role and Predictive Value of Human epididymis secretory protein 4 (HE4) and the Innate Immunity of the Oral Cavity and Respiratory Tract. Microorganisms. 2020 Nov 2;8(11):1718. doi: 10.3390/microorganisms8111718. PMID 33147871
- [Result] Nagata T, Yasuda Y, Ando M, Abe T, Katsuno T, Kato S, Tsuboi N, Matsuo S, Maruyama S. Clinical impact of kidney function on presepsin levels. PLoS One. 2015 Jun 1;10(6):e0129159. doi: 10.1371/journal.pone.0129159. eCollection 2015. PMID 26030716
- [Result] Ferrarese A, Frigo AC, Mion MM, Plebani M, Russo FP, Germani G, Gambato M, Cillo U, Cattelan A, Burra P, Senzolo M. Diagnostic and prognostic role of presepsin in patients with cirrhosis and bacterial infection. Clin Chem Lab Med. 2020 Oct 23;59(4):775-782. doi: 10.1515/cclm-2020-1212. Print 2021 Mar 26. PMID 33095752
- [Result] Zhang X, Liu D, Liu YN, Wang R, Xie LX. The accuracy of presepsin (sCD14-ST) for the diagnosis of sepsis in adults: a meta-analysis. Crit Care. 2015 Sep 11;19(1):323. doi: 10.1186/s13054-015-1032-4. PMID 26357898
- [Result] Memar MY, Baghi HB. Presepsin: A promising biomarker for the detection of bacterial infections. Biomed Pharmacother. 2019 Mar;111:649-656. doi: 10.1016/j.biopha.2018.12.124. Epub 2019 Jan 3. PMID 30611989